CLINICAL TRIAL: NCT05794373
Title: Education of Municipality-based Physiotherapists in Managing Disabling Low Back Pain - an Observational Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Spine Centre of Southern Denmark (Other)
Responsible Party: Principal Investigator, Thorvaldur Skuli Palsson, Head of research,, Aalborg University Hospital
Other Study IDs: Back pain in Municipalities
Record Dates: First submitted 2023-02-03; First posted 2023-04-03 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain; Rehabilitation; Physiotherapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Education group: Patients in this group undergo rehabilitation for back pain in a municipality setting with physiotherapists before the physiotherapists have participated in an educational intervention
  Interventions: Procedure: Standard physiotherapy for low back pain in a municipality setting
- Post-Education group: Patients in this group undergo rehabilitation for back pain in a municipality setting with physiotherapists after they have participated in an educational intervention
  Interventions: Procedure: Standard physiotherapy for low back pain in a municipality setting

INTERVENTIONS:
Procedure: Standard physiotherapy for low back pain in a municipality setting — Patients (N=100) referred to a municipality-based rehabilitation for low back pain are included. The physiotherapists choose the rehabilitation strategy based on what they consider relevant for the patients. After the first 100 patients have been discharged from municipality care, the physiotherapists will participate in an educational intervention (12 sessions) focusing on the management of low back pain within a multidimensional framework. In the educational intervention, the participants will learn how to identify the presence of unhelpful thoughts and emotions and how to address these as part of the intervention. The course will thus be a mix of theoretical and practical teaching, including case supervision and feedback. Following the educational intervention, an additional 100 patients referred to the rehabilitation program will be included. The intervention is aimed at the physiotherapists where the patients will receive the best available care, before or after the intervention.

SUMMARY:
A consistent theme in the modern-day healthcare system is the difficulty of transferring research knowledge into clinical practice. Recently, it has been pointed out that this is a barrier for providing care that is evidence-based which may partly explain the growing burden of low back pain.

Low back pain, as all other musculoskeletal pain conditions is multidimensional where biomedical and psychological factors need to be accounted for, as well as the patient's social context. From the healthcare provider perspective, this requires skills that often goes beyond the basic training where clinicians need to be able to assess and manage the multiple domains in a patient-centered manner.

In Denmark, people living with disabling low back pain can be referred to a municipality-based rehabilitation program. This study seeks to investigate whether providing physiotherapists an evidence-based educational course on the management of low back pain will change patient-related outcomes. Likewise, we will investigate potential barriers and facilitators for implementing the skills the physiotherapists acquire in clinical practice.

If the project shows a favorable effect, it will allow for upscaling the intervention within and across municipalities. Moreover, a positive outcome may provide indications of what type of continuing education resources should be made available to help clinicians better manage complicated low back pain problems.

DETAILED DESCRIPTION:
Schedule of procedures and assessments

1. All participating physiotherapists will recruit eligible patients (N=100) who are asked to fill out project-specific questionnaires (see procedures) at the start and at the end of the rehabilitation program.

2. The participating physiotherapists will undergo a 13-day educational intervention (see description below under intervention) focusing on management of low back pain within an individualized multidimensional framework.

3. Point 1 is repeated on an additional 100 patients who undergo rehabilitation after the physiotherapists have completed the course

4. Participating physiotherapists will be evaluated on the background of a competency checklist which is scored by clinical supervisors connected to the study. The checklist will be scored after watching a video recording of a patient consultation performed by the physiotherapist in focus. The checklist covers 6 domains: Subjective and objective assessment, cognitive-functional therapy intervention, style of communication, patient's unhelpful pain behavior, and an overall assessment

5. Physiotherapists who demonstrate high and low competency (as determined by the evaluation of competency, point 4) are invited to participate in a semi-structured interview. The interview will explore the physiotherapists' experience of changes in management (if any) after the educational intervention. This includes challenges, barriers and facilitating factors.

Intervention All procedures will be based on the physiotherapists assessment where individual needs and goals are embedded into the rehabilitation. The project will investigate whether priorities within assessment and choice of management change after the educational intervention. The educational program for the physiotherapists will run over 13 days and is divided into 3 overlapping modules.

Module 1 (5 days) - Evidence-based theory The module will focus on theoretical and practical aspects of the management of patients with back pain within a multidimensional framework. This includes differential diagnostics, social medicine measures, communication training with a focus on motivational interview and management of patients with dominant cognitive and emotional factors.

An evidence-based overview of contributing factors to the pain experience will be addressed including lifestyle, emotions, cognitions, response to pain including protective movement strategies, co-morbidity, activity level, physical/mental stress, patho-anatomy, nervous system sensitivity and social factors.

Module 2 (3 days) - Masterclass Masterclass in where two experienced clinicians from the project group will demonstrate patient examinations and management of complex low back patients. The purpose is to help the participants gain insight into clinical application of relevant multi-dimensional management of disabling low back pain. These demonstrations provide the platform for the following module 3.

Module 3 (5 days) - Clinical supervision In the supervision sessions the participants receive training/guidance in integrating the theoretical and practical skills from the previous modules. Feedback/evaluation from supervisors ensures that the participants adapt a multi-dimensional perspective in their patient management. Competency is tested here

ELIGIBILITY:
The following criteria apply for the patients entering the study

Inclusion Criteria:

* referred to municipality care from the Spine Clinic of Southern Denmark
* Between 18-65 years
* Speaks and comprehends Danish
* A score over 40 on the Orebro Musculoskeletal Pain Questionnaire
* Low back pain as dominating cause for referral

Exclusion Criteria:

* A current diagnosis of psychiatric illness that precludes participation in rehabilitation
* A neurologic disorder or other disease that may affect the ability to participate in a municipality based rehabilitation program
* A neurological deficits related with radiographically confirmed lumbar spinal stenosis or radicular pain correlating with the clinical presentation
* Recent (within 6 months) history of a stabilizing operation of the low back

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physiotherapists working in a municpality setting (N=25) in the region of southern Denmark. Minimum one year clinical experience in working with spine-related disorders
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disability | At baseline and 3 months after starting rehabilitation
  Change in disability measured on the Roland Morris Disability Questionnaire between baseline and follow up.
  Questionnaire designed to capture disability in low back pain patients (0-24 where 0 = no loss of function and 24 = complete loss of function)

SECONDARY OUTCOMES:
Pain intensity | At baseline and 3 months after starting rehabilitation
  Change in pain intensity between baseline and follow-up on a numeric rating scale (NRS: 0-10) Pain intensity scores (Average, best and worst). 0 is no pain; 10 is worst pain imaginable
Emotional and cognitive functioning | At baseline and 3 months after starting rehabilitation
  Orebro Musculoskeletal Pain Questionnaire. The questionnaire captures psychological and emotional factors in musculoskeletal pain. In the study, the questionnaire is used as a screening tool to determine eligibility. The score ranges from 4-210 where a higher score indicates greater loss of function related to cognitive or emotional factors. A cut-off score for entering the study is set at 40
Sick leave from work | At baseline and 3 months after starting rehabilitation
  Patients indicate whether they are on sick leave. If yes, whether they are on full sick leave or have reduced work capacity (indicated in hours per week) or normal work capacity
Patient Assessment of Transitions in Healthcare | 3 months after starting rehabilitation
  The participants evaluate the quality and coherence in management of their condition across sectors by indicate to what degree a range of statements on a 5 point Likert scales ranged from 'strongly disagree' to 'strongly agree'. The total score does not indicate a better or worse outcome but simply to what degree the statements apply to the patients' transition through the healthchare system

OTHER OUTCOMES:
Checklist to determine the competency of clinicians | Up to 24 weeks after the project period has ended
  Participating physiotherapists will be evaluated on the background of a competency checklist which is filled out by two of the study's assessors. The checklist will be filled out after watching af video recording of a patient consultation performed by the physiotherapist in focus. The checklist covers 6 domains: Subjective and objective assessment, cognitive-functional therapy intervention, style of communication, patient's unhelpful pain behavior, and an overall assessment. On each domain the participants are evaluated on the basis of whether they are no competent, developing their competency or competent.
  The assessors will be be blind to whether the video is recorded prior to or after the participating physiotherapists have been through the educational intervention
Barriers and facilitators for implementing new knowledge in clinical practice - qualitative interview | Up to 24 weeks after the project period has ended
  Physiotherapists who have participated in the educational intervention are invited to participate in a semistructured interview. The focus of the interview will be on the physiotherapists' experience of changes in management (if any) after the educational intervention. This includes challenges, barriers and facilitating factors

CONTACTS AND LOCATIONS:
Overall Officials: Thorvaldur S Palsson, PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Spine Center of Southern Denmark, Middelfart, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT05794373/Prot_SAP_000.pdf